CLINICAL TRIAL: NCT05208541
Title: Advancing Dignity, Health, and Optimism in Connection With Long Acting Injectables
Acronym: ADHOC-LA
Status: Recruiting | Type: Observational
Sponsor: Mazonson & Santas Inc. (Industry)
Collaborators: AIDS Healthcare Foundation (Other); Be Well Medical Center (Unknown); Central Texas Clinical Research (Unknown); The Crofoot Research Center, Inc. (Industry); Gary J. Richmond, MD (Unknown); Hennepin County Medical Center, Minneapolis (Other); Icahn School of Medicine at Mount Sinai (Other); Infectious Diseases Association of Central VA (Unknown); KC Care Health Center (Other); Long Beach Education and Research Consultants (Unknown); Mills Clinical Research (Industry); North Texas Infectious Disease Consultants (Unknown); Felizarta, Franco, M.D. (Individual); Prism Health North Texas (Other); Texas Centers for Infectious Disease Associates (Unknown); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ADHOC-LA 1001
Record Dates: First submitted 2021-12-21; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: HIV
Keywords: HIV; PLWH; Long Acting Injectable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ADHOC-LA is an observational study of people living with HIV who either are taking, or have taken, a long-acting injectable therapy to manage their HIV. Data from this study will be used to research the ways in which HIV impacts the lives of these patients.

DETAILED DESCRIPTION:
ADHOC-LA is an observational study that uses an online questionnaire to collect data on adults living with HIV who are currently taking, or have previously taken, long-acting injectable therapy to manage their HIV. The questionnaire includes information on sociodemographic factors, activities and interests, HIV diagnosis and status, health care use and satisfaction, antiretroviral therapy, comorbid medical conditions, health and well-being, substance use, and sexual practices.

ELIGIBILITY:
Eligibility Criteria:

1. Have an HIV-1 infection
2. a) Currently take a long-acting injectable therapy for HIV supplied by ViiV as part of a ViiV-sponsored, long-acting injectables therapy trial (LATTE-2, ATLAS-2M, CUSTOMIZE, POLAR, FLAIR, or SOLAR), or

   b) Currently take a long-acting injectable therapy for HIV prescribed by their provider, not in conjunction with a ViiV-sponsored clinical trial, or

   c) No longer taking long-acting injectable therapy for HIV, but previously received three or more injections of long-acting injectable therapy, either:
   * Supplied by ViiV as part of a ViiV-sponsored, long-acting injectables therapy trial (LATTE-2, ATLAS-2M, CUSTOMIZE, POLAR, FLAIR, or SOLAR), or
   * Prescribed by their provider, unrelated to a ViiV-sponsored clinical trial.
3. Age 18 or above
4. Have no known acute medical problem requiring immediate inpatient treatment
5. Able to read and write in English
6. Able and willing to provide online informed consent and to complete the online profile
7. Not currently enrolled in another clinical trial in which the participant is receiving a long-acting injectable therapy for HIV.

Participants who meet the eligibility criteria but are still receiving ViiV-supplied drug may enroll in the registry, but will not begin the online questionnaire until they are rolled off of ViiV-supplied long-acting injectable therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People over the age of 18 with an HIV-1 infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Baseline
  Measured using the Three-Item Loneliness Scale. This scale is comprised of 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. The scale range of each response item is 1-3. The total score ranges from 3-9 with higher total scores indicating a higher level of perceived loneliness.
Loneliness | Through study completion, an average of 12 months
  Measured using the Three-Item Loneliness Scale. This scale is comprised of 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. The scale range of each response item is 1-3. The total score ranges from 3-9 with higher total scores indicating a higher level of perceived loneliness.
Quality of life measurement | Baseline
  Measured using the PozQoL. PozQoL is a short 13-question scale assessing quality of life among people living with HIV. The scale includes four subscales: health concerns, psychological, social and functional. The scale range of each response item is 1-5. The total score is the average of all response items ranges from 1-5 with higher total scores indicating higher quality of life.
Quality of life measurement | Through study completion, an average of 12 months
  Measured using the PozQoL. PozQoL is a short 13-question scale assessing quality of life among people living with HIV. The scale includes four subscales: health concerns, psychological, social and functional. The scale range of each response item is 1-5. The total score is the average of all response items ranges from 1-5 with higher total scores indicating higher quality of life.
Cognitive function | Baseline
  Measured using the Functional Assessment of HIV Infection (FAHI Cognition). The FAHI Cognition subscale is used to create a standardized score to assess outcome. The scale range of each response is 0-4. The total score has a range of 0-12 with higher total scores indicating a higher cognitive functioning.
Cognitive function | Through study completion, an average of 12 months
  Measured using the Functional Assessment of HIV Infection (FAHI Cognition). The FAHI Cognition subscale is used to create a standardized score to assess outcome. The scale range of each response is 0-4. The total score has a range of 0-12 with higher total scores indicating a higher cognitive functioning.
Social well-being | Baseline
  Measured using the Functional Assessment of HIV Infection (FAHI). The FAHI Social Well-being subscale will be used to create a standardized score to assess outcome. The scale range of each response is 0-4. The total score has a range of 0-32 with higher total scores indicating better social well-being.
Social well-being | Through study completion, an average of 12 months
  Measured using the Functional Assessment of HIV Infection (FAHI). The FAHI Social Well-being subscale will be used to create a standardized score to assess outcome. The scale range of each response is 0-4. The total score has a range of 0-32 with higher total scores indicating better social well-being.
Depression | Baseline
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). The scale range of each response item is 0-3. The total score for depression has a range from 0-6 with higher scores indicating positive for depression.
Depression | Through study completion, an average of 12 months
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). The scale range of each response item is 0-3. The total score for depression has a range from 0-6 with higher scores indicating positive for depression.
Anxiety | Baseline
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). The scale range of each response item is 0-3. The total score for anxiety has a range from 0-6 with higher scores indicating positive for generalized anxiety.
Anxiety | Through study completion, an average of 12 months
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). The scale range of each response item is 0-3. The total score for anxiety has a range from 0-6 with higher scores indicating positive for generalized anxiety.
Sleep quality | Baseline
  Measured using The Medical Outcomes Study Sleep Scale (MOS-SS). MOS-SS includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. The scale range of each response item is 0-100. The total score is the average of all response items and has a range of 0-100 with higher scores indicating poorer sleep quality.
Sleep quality | Through study completion, an average of 12 months
  Measured using The Medical Outcomes Study Sleep Scale (MOS-SS). MOS-SS includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. The scale range of each response item is 0-100. The total score is the average of all response items and has a range of 0-100 with higher scores indicating poorer sleep quality.
Alcohol use | Baseline
  Measured using the Alcohol Use Disorder Identification Test (AUDIT-C). The AUDIT-C is a 3-item screening survey that can help identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The scale range of each response item is 0-4. The total score has a range of 0-12 with a higher score indicating more hazardous drinking behavior.
Alcohol use | Through study completion, an average of 12 months
  Measured using the Alcohol Use Disorder Identification Test (AUDIT-C). The AUDIT-C is a 3-item screening survey that can help identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The scale range of each response item is 0-4. The total score has a range of 0-12 with a higher score indicating more hazardous drinking behavior.
Internalized stigma | Baseline
  Measured using the Internalized AIDS-Related Stigma scale (IAS). IAS is a six-item scale designed to measure the construct of internalized stigma. The scale range of each response item is 0-1. The total score has a range of 0-6 with higher scores indicating more internalized stigma.
Internalized stigma | Through study completion, an average of 12 months
  Measured using the Internalized AIDS-Related Stigma scale (IAS). IAS is a six-item scale designed to measure the construct of internalized stigma. The scale range of each response item is 0-1. The total score has a range of 0-6 with higher scores indicating more internalized stigma.
Resilience | Baseline
  Measured using the Connor-Davidson Resilience Scale (CD-RISC 2). The CD-RISC contains two items and was developed as a measure of "bounce-back" and adaptability. The scale range of each response item is 0-8. The total score range is 0-16 with higher scores indicating higher resilience.
Resilience | Through study completion, an average of 12 months
  Measured using the Connor-Davidson Resilience Scale (CD-RISC 2). The CD-RISC contains two items and was developed as a measure of "bounce-back" and adaptability. The scale range of each response item is 0-8. The total score range is 0-16 with higher scores indicating higher resilience.
Interpersonal support | Baseline
  Measured using the Interpersonal Support Evaluation Checklist - 6 (ISEL-6). ISEL-6 is derived from the long form of the ISEL and contains 6 items that assess the perceived availability of social support. The scale range of each response item is 1-4. The total score range is 6-48 with higher scores indicating higher social support.
Interpersonal support | Through study completion, an average of 12 months
  Measured using the Interpersonal Support Evaluation Checklist - 6 (ISEL-6). ISEL-6 is derived from the long form of the ISEL and contains 6 items that assess the perceived availability of social support. The scale range of each response item is 1-4. The total score range is 6-48 with higher scores indicating higher social support.
Anti-HIV medication adherence | Baseline
  Measured using the brief adherence self-report questionnaire. This questionnaire asks participants how much of their anti-HIV medications they have taken over the past month (0 to 100%). Higher score indicates greater adherence to anti-HIV medication(s).
Anti-HIV medication adherence | Through study completion, an average of 12 months
  Measured using the brief adherence self-report questionnaire. This questionnaire asks participants how much of their anti-HIV medications they have taken over the past month (0 to 100%). Higher score indicates greater adherence to anti-HIV medication(s).
Frailty | Baseline
  Measured using the Frailty Index Elders (FIFE). FIFE is a 10-item instrument with scores ranging from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty.
Frailty | Through study completion, an average of 12 months
  Measured using the Frailty Index Elders (FIFE). FIFE is a 10-item instrument with scores ranging from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty.

OTHER OUTCOMES:
Sociodemographic Characteristics | Baseline
  Demographic characteristics including, but not limited to, age, sex, race, body weight, income, and education will be evaluated as potential predictors of inter- and intra-participant variability for patient-reported outcome measures.
Sociodemographic Characteristics | Through study completion, an average of 12 months
  Demographic characteristics including, but not limited to, age, sex, race, body weight, income, and education will be evaluated as potential predictors of inter- and intra-participant variability for patient-reported outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Mazonson & Santas Inc, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Undecided